CLINICAL TRIAL: NCT06020573
Title: Evaluation of Safety and Performance of Intraoperative Detection of Light Signals During Electrosurgical Breast Cancer Resection (ELINORE)
Brief Title: Evaluation of Safety and Performance of Intraoperative Detection of Light Signals During Electrosurgical Breast Cancer Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erbe Elektromedizin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 768/2022MP1
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Resection Margin
MeSH Terms: conditions — Breast Neoplasms; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intraoperative detection of light signals during electrosurgical breast cancer resection (Other): Participants undergo electrosurgical breast cancer resection while light signals are detected intraoperatively
  Interventions: Device: Clip-on electrode with fiber optics

INTERVENTIONS:
Device: Clip-on electrode with fiber optics — The device will be used for tumor resection of breast cancer and for the collection of optical data that could be ultimately used for providing additional information.

SUMMARY:
This monocentric early feasibility first in human study is intended to evaluate safety and performance of intraoperative detection of light signals during electrosurgical breast cancer resection.

In consequence the data should also be taken to adapt technical features according to the findings. The study results will be utilized to design and to calculate the sample size for future pivotal studies after finalizing this study and to adapt the technical features of the system and/ or device. In the future pivotal study, the effectiveness of method and the reduction in R1 resection rate will be assessed with the final goal to provide continuous or real-time information about the tissue type that is currently cut.

The primary endpoint for this first in human feasibility study is the percentage of patients with no serious adverse event related to the investigational device.

After signing the informed consent the doctor and research team will determine if the participant meets all requirements for this study. During the second visit (V2) they will receive the treatment procedure with the investigational medical device (IMD). The follow up visit (V3) will be performed up to 7 days after the treatment procedure at the day of discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient with primary invasive breast cancer (NST or NST with DCIS component, including endocrine pretreatment according to standard of care therapy at the study site)
2. Solid tumor size ≥ 15 mm at screening, on sonography imaging
3. Breast conserving surgery
4. ≥ 18 years of age
5. Ability to provide written informed consent

Exclusion Criteria:

1. Neoadjuvant chemotherapy
2. Bilateral breast conserving surgery
3. Invasive lobular carcinoma, DCIS, LCIS
4. Suspicion of extensive DCIS component of NST tumor
5. Diagnosis of recurrent breast cancer
6. Previous radiotherapy
7. Patient is pregnant or lactating
8. Patient is wearing active implant (cardiac pacemaker, internal defibrillator, other active implant), passive implants (hip arthroplasties, tooth implants etc.) are allowed at the discretion of the principal investigator
9. According to physicians' assessment, patient is not able to follow study protocol (e.g., due to cognitive disease) or is not able to understand the nature, objectives, benefits, implications, risks and inconveniences of the clinical investigation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Safety, feasibility and performance | 11 days
  The primary endpoint for this first in human feasibility study is the percentage of patients with no serious adverse event related to the investigational device.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Hahn, Prof.Dr. Med., Principal Investigator — Department for Women's Health, Tuebingen, Germany
Locations (1):
- Department for Women's Health, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spether D, Scharpf M, Hennenlotter J, Schwentner C, Neugebauer A, Nussle D, Fischer K, Zappe H, Stenzl A, Fend F, Seifert A, Enderle M. Real-time tissue differentiation based on optical emission spectroscopy for guided electrosurgical tumor resection. Biomed Opt Express. 2015 Mar 24;6(4):1419-28. doi: 10.1364/BOE.6.001419. eCollection 2015 Apr 1. PMID 25909025